CLINICAL TRIAL: NCT02607371
Title: AF Patient Preferences Towards NOAC Versus VKA Treatment: a Patient Preference Study
Brief Title: Anticoagulation Preference by AF Patients Study
Acronym: PRiSMA-AF
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18242
Record Dates: First submitted 2015-08-27; First posted 2015-11-18 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation
Keywords: Patient treatment preference; Non-valvular Atrial Fibrillation; NOAC; VKA
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; edoxaban; apixaban; Dabigatran

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1 / VKA treatment: A sample of about 200 patients with nonvalvular atrial fibrillation who are treated with VKAs for at least three months at date of study inclusion
  Interventions: Other: VKAs
- Cohort 2 / NOAC treatment: A sample of about 200 patients with nonvalvular atrial fibrillation who are treated with NOACs for at least three months at date of study inclusion
  Interventions: Other: NOACs including Rivaroxaban (Xarelto, BAY59-7939); Other: Edoxaban; Other: Apixaban; Other: Dabigatran-etexilate

INTERVENTIONS:
Other: VKAs — VKA have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: Cohort 1 / VKA treatment
Other: NOACs including Rivaroxaban (Xarelto, BAY59-7939) — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: Cohort 2 / NOAC treatment
Other: Edoxaban — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: Cohort 2 / NOAC treatment
Other: Apixaban — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: Cohort 2 / NOAC treatment
Other: Dabigatran-etexilate — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: Cohort 2 / NOAC treatment

SUMMARY:
The main research question of this patient survey is to assess AF (Atrial Fibrillation) patients' preferences associated with different attributes which describe the different available anticoagulation treatment options (Vitamin K Antagonists [VKA] or New Oral Anticoagulants [NOACs] and, in case of NOACs, Apixaban, Dabigatran, Edoxaban or Rivaroxaban).

VKAs (Marcoumar®, Sintrom ®) will be grouped together and compared to Rivaroxaban.

DETAILED DESCRIPTION:
The objective of this study is to investigate the following research questions in a cross-sectional survey of German-speaking Swiss AF patients being treated either with a VKA or with a NOAC:

* Which attributes of a medication to prevent stroke do AF patients view as important?
* Do AF patients have a preference regarding the attributes of the medication options VKA or NOAC and, in case of NOACs, with regards to rivaroxaban attributes?
* Are there subgroups of AF patients whose preference for one of the medication options appears above or below average?
* What is the quality of life of Swiss German-speaking AF patients? Are there subgroups with differences in their quality of life (for example: subgroups of patients with different CHA2DS2-VASc scores)?
* Which burden do German-speaking Swiss AF patients experience in association with their anticoagulation therapy? Are there differences in the burden of treatment (ACTS) between patients treated with VKA or with NOACs?

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for AF patients in both the NOAC and the VKA groups:

* Patients with a confirmed diagnosis of nonvalvular atrial fibrillation (persistent, paroxysmal, permanent),
* Age of at least 18 years at time of study inclusion,
* Generally willingness (informed consent) and ability to fill out a survey on satisfaction with treatment and quality of life, and to conduct a structured phone interview (approx. 20 - 30 min) in German language.

Additional inclusion criterion for Group 1 (NOAC):

* Continuous anticoagulation with either Apixaban, or Dabigatran or Rivaroxaban for prevention of Stroke & systemic embolism for at least the previous 3 months.

Additional inclusion criterion for Group 2 (VKA):

* Continuous anticoagulation with a VKA for prevention of Stroke & systemic embolism for at least the previous 3 months.

Exclusion Criteria:

Exclusion criteria for both groups:

* Participation in another study (clinical intervention / observational) within the 3 months prior to enrollment,
* Interruption of VKA/NOAC therapy of more than 2 weeks (bridging) within the prior 3 months or planned bridging in 4 weeks after study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in primary care / general outpatient practices and outpatient clinics in German-speaking Switzerland.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
AF patients'preferences towards anticoagulation treatment with either VKAs or NOACs measured with a DCE (discrete choice experiment) design in a phone interview | up to 4 weeks
  * DCE is based on the following attributes /attribute levels:
  * Frequency of intake (once/twice daily),
  * Need of INR monitoring/dose adjustment (yes/no),
  * Need of bridging (yes/no),
  * Interactions with food/drugs (yes/no),
  * Distance to treating physician (1km or 15km).

SECONDARY OUTCOMES:
Burden associated with anticoagulation treatment measured by the questionnaire ACTS | Baseline
Health-related quality of life measured by the SF-12 questionnaire | up to 4 weeks
  Variables: Physical/psychological domain according to SF-12 questionnaire
Assessment of factors that may be associated with AF patients preferences towards a specific anticoagulation treatment: preferred anticoagulation treatment (agent) | up to 4 weeks
Assessment of factors that may be associated with AF patients preferences towards a specific anticoagulation treatment: HrQoL as defined by the SF-12 score | up to 4 weeks
Assessment of factors that may be associated with AF patients preferences towards a specific anticoagulation treatment: AF symptoms as measured by the EHRA | up to 4 weeks
Assessment of factors that may be associated with AF patients preferences towards a specific anticoagulation treatment: TTR (for VKA patients only) | up to 4 weeks
Assessment of factors that may be associated with AF patients preferences towards a specific anticoagulation treatment: Age | up to 4 weeks
Assessment of factors that may be associated with AF patients preferences towards a specific anticoagulation treatment: Gender | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Switzerland